CLINICAL TRIAL: NCT06184360
Title: Real-world Evaluation of BEOVU (Brolucizumab) Effectiveness and Durability for Treatment of Neovascular (Wet) Age-related Macular Degeneration (AMD)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258A2014
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Neovascular (Wet) Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Treatment-Experienced
- Treatment-Naive

SUMMARY:
This was a retrospective, observational cohort study. Data were analyzed from the Intelligent Research in Sight (IRIS) registry from October 8, 2019, through November 26, 2021, with a follow-up period of 12 months following the first brolucizumab injection (index date).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old at the time of their first (index) injection of brolucizumab.
* Had documented neovascular age-related macular degeneration (nAMD) on or within 3 years before the index injection.
* Used only brolucizumab for at least 12 months (± 45 days) after the index injection, with at least 1 brolucizumab injection given within the first 6 months after the index injection and at least 1 additional brolucizumab injection given at 6-12 months after the index injection.

Exclusion Criteria:

* Had received any other anti-VEGF agent between the index injection and 12-month follow-up.
* Lacked information about the laterality of disease at the time of the index injection.
* Lacked visual acuity assessments on or within 30 days before the index injection or at 6, 9, and 12 months after the index injection (all of the latter ± 45 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 2079 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Change in Best Recorded Visual Acuity, Stratified by Prior Treatment Status | Baseline up to 12 months
Change in Injection Interval at 12 Months of Brolucizumab Treatment Compared with Prior Anti-vascular Endothelial Growth Factor (VEGF) Treatment | Baseline up to 12 months
Number of eyes with adverse events | Baseline up to 12 months
Time to adverse event | Baseline up to 12 months
Number of brolucizumab injections prior to adverse event | Baseline up to 12 months

SECONDARY OUTCOMES:
Brolucizumab Injection Interval and Interval Extension, Stratified by Pre-Switch Interval | Baseline up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States